CLINICAL TRIAL: NCT05015205
Title: Effects of Muscle Energy Technique and Postural Correction Exercises in Lordotic Females Wearing High Heels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/RCRS/18/1003
Record Dates: First submitted 2021-08-10; First posted 2021-08-20 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Lordosis; Low Back Pain
Keywords: Lordosis; METs; Postural Correction Exercise
MeSH Terms: conditions — Lordosis; Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MET Group (Experimental): Post isometric relaxation technique MET was applied in two muscle groups; Lumbar Extensors (Erector Spinae) and Hip Flexors (Iliopsoas). The exercises were performed 3 times per week for 4 weeks.
  Interventions: Other: Muscle Energy Technique
- Control Group (Experimental): Postural Correction Exercises was applied to one group. Exercises performed included stretching and strengthening exercises. The exercises were performed 3 times per week for 4 weeks.
  Interventions: Other: Postural Correction Exercises

INTERVENTIONS:
Other: Muscle Energy Technique — Post isometric relaxation technique MET was applied in two muscle groups; Lumbar Extensors (Erector Spinae) and Hip Flexors (Iliopsoas). The muscle was positioned in position and patient was asked to apply 20% force isometrically and hold the isometric contractions for 7-10 seconds. Then the patient was asked to relax for about seconds. On exhalation, therapist takes muscle to new restriction barrier. Hold this position for 30 seconds at the end barrier as an end-stretch with 3 repetitions.
  Arms: MET Group
Other: Postural Correction Exercises — : Postural Correction Exercises was applied to one group. Exercises performed included stretching and strengthening exercises. Hip flexors and back extensors were stretched while hip extensors and abdominals were strengthened. Seated hip flexion used to stretch back extensors while lunge position used to stretch hip flexors. The abdominals were strengthened by using curl up exercises while hip extensors were strengthened by resisted contractions in prone lying.
  Arms: Control Group

SUMMARY:
The key purpose was to determine the effects of Muscle Energy Technique (MET) and Postural Correction Exercises on low back pain in females wearing high heels.

To determine the effects of muscle energy technique & postural correction exercises in reducing pain, anterior pelvic tilt angle and increasing lumbar range of motion in subjects with chronic low back pain due to lordotic posture in females wearing high heels.

DETAILED DESCRIPTION:
Body segments can be defined as the suitable posture positions. Body segments are placed in a way that center of gravity of each segment lies vertically. By this appropriate alignment, instead of excessive muscular activity, stability can be achieved by the body by the use of bone structures and ligament. Hence, in this way body structures experience the decreased tension. Besides the cosmetic effects of high heels, high heels results in increased risk of fall, fracture of bones particularly bones lower extremity, and also the change in normal kinematics of lower limb especially knee joint, and altered weight bearing on medial and longitudinal arches of foot. High heels change the line of gravity and posture of the body. Use of high heels change the posture which is compensated by the changes in different segments of the body like increased planter flexion of ankle as well as the displacements of the trunk and posterior pelvic tilting. The whole body mechanics gets affected in females wearing high heels. The center of gravity get disturbed with the use of high heel shoes. In body alignment, pelvis is known to have key importance. Any alteration in neutral position of pelvis leads to the compensatory altered movements in different regions, while, the segment which is considered to be the most effect is lumber spine.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-45 years
2. Low back pain of no more than 12 weeks duration in lordotic females wearing high heel shoes.
3. Females wearing 4 to 5 inches high heel shoes 6 hour per day.
4. Increased lumbosacral angle
5. An initial ODI score of 20 % to 60 %.
6. Localized pain in lumbar spine with no radiating pain towards buttocks, hips or legs.

Exclusion Criteria:

1. Any red flags (tumor, fracture, metabolic diseases, rheumatoid arthritis, osteoporosis, resting blood pressure greater than 140/90 mmHg, prolonged history of steroid use, etc)
2. Presented with involvement of nerve compression symptoms like radiating pain, change in normal sensory sensations with significant muscle weakness, or hypo reflexia or hyper reflexia.
3. Presented with a diagnosis of Lumbar spinal stenosis.
4. Presented with a diagnosis of Lumbar spinal spondylolisthesis.
5. Prior surgery to the lumbar region.
6. Patients who are already receiving treatment.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Females wearing high heels
Enrollment: 28 (Actual)
Dates: Start 2019-04-02 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | 3 months
  This is subjective instrument that is widely used in clinical settings. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").
Disability Index (DI) | 3 months
  This is subjective instrument that is widely used in clinical settings. 0% to 20%: minimal disability: The patient can cope with most living activities. Usually no treatment is indicated apart from advice on lifting sitting and exercise. 21%-40%: moderate disability: The patient experiences more pain and difficulty with sitting, lifting and standing. Travel and social life are more difficult and they may be disabled from work. Personal care, sexual activity and sleeping are not grossly affected and the patient can usually be managed by conservative means. 41%-60%: severe disability: Pain remains the main problem in this group but activities of daily living are affected. These patients require a detailed investigation. 61%-80%: crippled: Back pain impinges on all aspects of the patient's life. Positive intervention is required. 81%-100%: These patients are either bed-bound or exaggerating their symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Nosheen Manzoor, MS, Principal Investigator — Riphah International University
Locations (1):
- Nosheen Manzoor, Faisalābad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No